CLINICAL TRIAL: NCT04624100
Title: Quality Control of Ventral Hernia Surgery in 21 Belgian Hospitals by Prospective Registration in Close Collaboration With the Danish Hernia Database.
Brief Title: Quality Control of Ventral Hernia Surgery by Prospective Registration
Status: Not yet recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Belgian Section for Abdominal Wall Surgery, section of the Royal Belgian Society for Surgery (Unknown)
Responsible Party: Principal Investigator, Marc Miserez, MD PhD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S62600
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Ventral Incisional Hernia
MeSH Terms: interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- All consecutive patients with primary ventral or incisional hernia
  Interventions: Procedure: Hernia repair

INTERVENTIONS:
Procedure: Hernia repair — Primary or mesh repair of primary ventral or incisional hernia

SUMMARY:
Quality Control of ventral hernia surgery in 21 Belgian hospitals by prospective registration in close collaboration with the Danish Hernia Database.

ELIGIBILITY:
Inclusion criteria

* Consecutively all patients with an elective or emergency repair of every ventral/incisional hernia (including parastomal hernia)
* Male and female
* 18 years or older
* Operated of supervised by a participating surgeon (participating in this study is not necessarily by a whole surgical department of one of the 18 participating Belgian hospitals, but by specific surgeons)
* Elective and emergency surgery
* Signed informed consent form

Exclusion criteria

* Younger than 18 years
* Not operated or supervised by participating surgeon
* Pregnant at inclusion in the registry
* No signed informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing primary ventral/incisional hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Reoperation | through study completion, an average of 2 years
  reoperation and readmission rate for (mesh-related) complications or recurrence related) complications or recurrence reoperation and readmission rate for (mesh related) complications or recurrence reoperation and readmission rate for (mesh related) complications or recurrence reoperation and readmission rate for (mesh related) complications or recurrence reoperation and readmission rate for (mesh related) complications or recurrence reoperation and readmission rate for (mesh related) complications or recurrence reoperation and readmission rate for (mesh-related) complications or recurrence